CLINICAL TRIAL: NCT00560677
Title: Schizophrenia and PTSD Project: Health, Interventions, and Risk/Resilience Evaluation
Brief Title: Schizophrenia and PTSD Project: Health, Interventions, and Risk/Resilience Evaluation(SAPPHIRE Study)
Acronym: SAPPHIRE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Durham VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: VA IRB# 01175; VA IRB# 01175
Record Dates: First submitted 2007-11-19; First posted 2007-11-20 (Estimated); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Schizophrenia; PTSD
Keywords: Schizophrenia; PTSD; Cognition
MeSH Terms: conditions — Schizophrenia; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum and cells collected.
Oversight: Data Monitoring Committee: No

SUMMARY:
We propose to establish a database characterizing the presence or absence of comorbid PTSD in veterans with schizophrenia or schizoaffective disorder (SAD) receiving services at the Durham VA Medical Center. In addition to the evaluation of PTSD symptoms in veterans with schizophrenia or SAD, this database will facilitate the investigation of a number of additional specific research questions relevant to veterans with psychotic disorders.

DETAILED DESCRIPTION:
See brief summary

ELIGIBILITY:
Inclusion Criteria:

1. 18-72 years of age, any ethnic group, either sex.
2. Diagnostic and Statistical Manual, Fourth Edition (DSM-IV) diagnosis of schizophrenia or schizoaffective disorder.
3. Ability to fully participate in the informed consent process, or have a legal guardian able to participate in the informed consent process.

Exclusion Criteria:

1. Unstable current medical or neurological illness.
2. Significant suicidal or homicidal ideation.
3. Pregnant women or women who could be pregnant.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veterans with schizophrenia or schizoaffective disorder.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2007-03; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Brief Assessment of Cognition in Schizophrenia (BACS) | Visit 1
  The Brief Assessment of Cognition in Schizophrenia (BACS) includes brief assessments of executive functions, verbal fluency, attention, verbal memory, working memory and motor speed. Z-scores are calculated from composite scores. Higher z-scores are indicative of better cognitive performance, lower z-scores are indicative of lower cognitive performance. Range of z-scores anticipated to be between -3 and 3.

CONTACTS AND LOCATIONS:
Overall Officials: Christine E Marx, MD, MA, Principal Investigator — Durham VAMC
Locations (1):
- Durham VAMC, Durham, North Carolina, United States